CLINICAL TRIAL: NCT05597410
Title: Shanghai At Risk for Alzheimer's Disease: a Cohort Study
Acronym: SHARAD
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHARAD-01
Record Dates: First submitted 2022-10-12; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease; Dementia; Neurodegenerative Diseases; Cognitive Impairment; Neurocognitive Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases; Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (3-4 ml) of all participants will be collected at baseline and stored at -80°C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cohort study is to estimate the incidence of AD in the first-degree relatives of patients with AD. The main questions it aims to answer are:

* cognitive changes of subjects at high risk of AD as ageing;
* environmental and behavioral factors affecting AD incidence.

DETAILED DESCRIPTION:
This study is a prospective cohort study focusing on the first-degree relatives of patients with Alzheimer's disease (AD). Multiple methods including the neuropsychiatric assessment battery, magnetic resonance imaging (MRI) and fluid biomarkers (blood and urine) are used to estimate the longitudinal changes of the participants at high risk of AD. Besides, a structured questionnaire is designed to investigate how environmental, behavioral and other factors influence the incidence of AD. This study is of great significance in establishing novel guidelines for the prevention and treatment of dementia suitable for Chinese population, and for clinicians to predict the risk of AD in first-degree relatives.

ELIGIBILITY:
Inclusion Criteria:

1. the AD diagnostic criteria of probands meet the 2011 National Institute on Aging - Alzheimer's Association framework, and participants are the first-degree relatives (including parents, children and siblings of the same father and mother) of the proband;
2. not patients with dementia;
3. ≥ 50 years, males and females;
4. subjects have lived in Shanghai for more than 1 year and have no plan to move out of Shanghai within 5 years;
5. subjects are able to complete investigation, physical examination, imaging examination and biological specimen collection.

Exclusion criteria:

Individuals will be excluded if they have:

1. other diseases which could cause cognitive decline, e.g. cerebrovascular diseases, Creutzfeldt-Jakob disease and Parkinsons disease;
2. history of psychological disorders (according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition);
3. uncorrectable visual or auditory impairment that hampers the completion of related examination.
4. pre-menopausal women will also be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is the first-degree, cognition-preserved relatives (including parents, children and siblings of the same father and mother) of patients with AD
Sampling Method: Non-Probability Sample
Enrollment: 3418 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of cognitive impairment at 5 years | 5 years
  Number of participants who covert to AD or mild cognitive impairment (MCI) will be recorded to calculate the incidence.

SECONDARY OUTCOMES:
Change From Baseline in Mini-Mental State Examination (MMSE) at 5 years | 5 years
  MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
Change From Baseline in Montreal cognitive assessment-Basic (MoCA) at 5 years | 5 years
  MoCA is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
Change From Baseline in Boston naming test (BNT) at 5 years | 5 years
  MoCA is a screening instrument used to assess object naming function. The total score ranges from 0 to 30, with lower scores indicating greater disease severity.
Change From Baseline in the auditory verbal learning test (AVLT) at 5 years | 5 years
  AVLT is a screening instrument used to assess the function of memory. The score in long-term memory (N5) ranges from 0 to 12, with lower scores indicating greater disease severity.
Change From Baseline in trail making test (TMT) at 5 years | 5 years
  AVLT is a screening instrument used to assess the executive function. Time consumed is recorded as the result, with higher scores indicating greater disease severity.
Change From Baseline in Geriatric Depression Scale (GDS) at 5 years | 5 years
  GDS is a neuropsychological scale used to assess the level of depression. The total score ranges from 0 to 30, with higher scores indicating greater disease severity.
Change From multi-modal MRI neuroimaging at 5 years | 5 years
  Evaluation of multimodal MRI, including high-resolution structural T1 imaging, functional MRI, diffusion tensor imaging and quantitative susceptibility mapping.

OTHER OUTCOMES:
Change From Baseline in Blood concentration of Phosphorylated Tau (p-tau) at 5 years | 5 years
  Blood p-tau 181 and p-tau 217 at baseline will be tested. The higher blood p-tau is a strong predictor for AD.
Change From Baseline in Blood Concentration of Amyloid β (Aβ) at 5 years | 5 years
  Blood Aβ40 and Aβ42 at baseline will be tested. The decreased blood Aβ42/40 ratio is a strong predictor for AD.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, MD, PhD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cannon-Albright LA, Foster NL, Schliep K, Farnham JM, Teerlink CC, Kaddas H, Tschanz J, Corcoran C, Kauwe JSK. Relative risk for Alzheimer disease based on complete family history. Neurology. 2019 Apr 9;92(15):e1745-e1753. doi: 10.1212/WNL.0000000000007231. Epub 2019 Mar 13. PMID 30867271